CLINICAL TRIAL: NCT02958358
Title: Evaluation of FDG Uptake and Pulmonary Perfusion by Positron Emission Tomography in Patients With Pulmonary Arterial Hypertension Before and After Treatment With Ambrisentan
Brief Title: FDG Uptake and Lung Blood Flow in PAH Before and After Treatment With Ambrisentan
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to recruit subjects
Sponsor: Robert Scott Harris, M.D. (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Robert Scott Harris, M.D., Associate Physician, Massachusetts General Hospital, Associate Professor, Harvard Medical School, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013P002592
Record Dates: First submitted 2015-04-06; First posted 2016-11-08 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary hypertension; ambrisentan; PET imaging; CT/PET
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary Hypertension (Experimental): Patients with Group I pulmonary arterial hypertension to undergo CT imaging, functional PET imaging before and after 3 months of treatment with ambrisentan
  Interventions: Other: CT imaging, functional PET imaging

INTERVENTIONS:
Other: CT imaging, functional PET imaging — Physiology study using CT and functional PET imaging with 13NN and FDG as radiotracers; images obtained before and 3 months after treatment with ambrisentan.

SUMMARY:
The investigators are doing this research study to find out how blood flow changes in the lungs of people with pulmonary hypertension before and after treatment with ambrisentan (sold under the brand name Letairis). The investigators hope that knowing about these differences will help us to better understand pulmonary hypertension and find new ways to diagnose it earlier.

DETAILED DESCRIPTION:
The overall goal of this study is to evaluate lung, large vessel, and right ventricular glucose uptake rate using 18FDG PET and distribution of pulmonary perfusion using 13NN PET in patients with pulmonary hypertension before and after treatment with ambrisentan. The investigators propose a pilot study of patients with Group I PAH. The investigators plan to complete this pilot study with 5 patients (projected enrollment of 8 to allow for drop-out rate). Taken together, the studies above demonstrate that FDG-PET can be used to detect changes associated with PAH, and to monitor response to therapy. FDG-PET is a widely available technology, and is firmly established in the field of clinical oncology. Ambrisentan is an endothelin receptor antagonist that is FDA-approved to treat patients with pulmonary arterial hypertension. Patients will be eligible for participation in this study if they have already made a decision to start treatment with ambrisentan for pulmonary hypertension. The investigators propose a physiologic study of patients who will already have made a decision to start ambrisentan therapy. Participation in the study will not alter or affect participants decisions regarding treatment.

Prior human studies evaluating response to PH-specific therapies focused only on the right ventricle. Oikawa et al. looked at the RV uptake in patients with PH and evaluated them before and after treatment with epoprostenol. Fang and colleagues used FDG-SPECT evaluate FDG uptake in the RV of patients with IPAH and PH before and after treatment with sildenafil. Both of those studies used SUV (specific uptake variable). The investigators propose to focus on the lung and the RV uptake rate (Ki) in order to provide a more robust analysis of the metabolic changes that underlie the development of pulmonary hypertension both in the right ventricle and the lung parenchyma, and to study the response to ambrisentan with FDG-PET.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female aged > or =18 years of age and < or =70 years.
2. Subject is diagnosed with pulmonary arterial hypertension (WHO Group I, by right heart catheterization (RHC), mean PA pressure > 25 and PCWP < 15) and planning to start therapy with ambrisentan, either as de-novo monotherapy or as part of combination therapy.
3. Subject has most recently undergone RHC within three months of entering the study.
4. If patient has been on PAH-specific therapy, the therapy (agent and dose) has been unchanged for at least three months.
5. The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
6. A signed and dated written informed consent is obtained from the subject.
7. Available to complete the study.
8. Able to fast for 6 hours prior to the study.
9. Able to lie flat and able to perform a 30 second breath hold.

Exclusion Criteria:

1. FEV1 and/or TLC < 70% predicted.
2. PCWP > 15 mm Hg.
3. Inability to perform the study (by primary MD or investigator assessment).
4. The subject is unable to perform the respiratory maneuvers necessary for the exam.
5. Subjects who have diabetes mellitus or glucose intolerance.
6. Subjects who have a known contraindication to ambrisentan.
7. Subjects who have a past or present disease, which as judged by the Investigators may affect the outcome of this study.
8. The subject has suspected history of drugs or alcohol abuse within the six months prior to the screening visit.
9. The subject is a woman of childbearing potential who is pregnant, seeking to become pregnant, or has a positive pregnancy test.
10. Subject with clinical instability in the judgment of the investigator, or hospitalization for progression of pulmonary hypertension or right heart failure in the three months prior to the study.
11. Subject with diagnosis of active tuberculosis, lung cancer, clinically overt bronchiectasis, allergic rhinitis, asthma, heart failure, ischemic heart disease, or COPD.
12. Subject that had a respiratory tract infection in the 4 weeks prior to the screening visit and throughout the duration of the study.
13. The subject has been exposed to a radiation dose over the past year that, when added to the radiation dose expected in this study, would exceed permissible yearly exposure as determined by the MGH radiation safety committee.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation of perfusion | One imaging visit lasting up to 3 hours
  Images will be generated with positron emission tomography that will be used to calculate the degree to which the blood flow in the lung is patchy rather than smooth. The statistical measure of this is called the coefficient of variation.

SECONDARY OUTCOMES:
FDG Uptake Rate (Ki) | One imaging visit lasting up to 3 hours
  To determine the FDG uptake (Ki) in the right ventricle, large pulmonary vessels, and pulmonary parenchyma to investigate the effect of treatment with ambrisentan on the RV, large vessel and pulmonary parenchyma 18FDG uptake rate and its relationship to invasive hemodynamic measurements, RV function by echo, functional class, 6MWT and serum NT-proBNP levels.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Harris, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
None obtained